CLINICAL TRIAL: NCT00146068
Title: Phase IV Double-Blind Randomized Study to Evaluate Safety and Efficacy of Interferon Beta-1a (Avonex) Plus Simvastatin (Zocor) Combination Therapy in Clinically Isolated Syndrome Suggestive of Multiple Sclerosis Over a One Year Period
Brief Title: EARLY IFNB-1a and Simvastatin Combination Therapy in Clinically Isolated Syndrome Suggestive of Multiple Sclerosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of North Carolina (Other)
Responsible Party: Silva Markovic-Plese, MD/Principal Investigator, UNC-Chapel Hill
Organization: University of North Carolina, Chapel Hill (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 04-NEUR-387
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Last update posted 2008-03-05 (Estimated); Status verified 2008-02

CONDITIONS: Multiple Sclerosis
Keywords: Clinically Isolated Syndrome
MeSH Terms: conditions — Multiple Sclerosis | interventions — Interferon beta-1a; Simvastatin

INTERVENTIONS:
Drug: Avonex/Zocor

SUMMARY:
The purpose of this study is to determine the safety, tolerability and efficacy of a combination therapy interferon beta-1a(Avonex) plus simvastatin (Zocor) vs. interferon beta-1a plus placebo in patients with clinically isolated syndrome suggestive of Multiple Sclerosis.

DETAILED DESCRIPTION:
Interferon beta-1a (IFNB-1a), a FDA approved therapy for relapsing-remitting (RR) MS has several mechanisms of action. It lowers proinflammatory cytokine production and inhibits antigen presentation by class II major histocompatibility complex (MHC) molecule. It also reduces metalloproteinase activity, which all lead to decreased migration of T-lymphocytes into the central nervous system (CNS), and subsequent inhibition of inflammatory lesion formation. We propose that combination therapy during early stages of the disease with second immunomodulatory agent that targets different steps in the pathogenesis of the disease may add to the effectiveness of IFNB-1a. IFNB-1a administered intramuscularly at 30 mg per week is particularly suitable for combination therapy due to its proven efficacy in Clinically Isolated Syndrome (CIS),favorable safety profile and low frequency of neutralizing antibodies (NABs) against IFNB-1a in comparison to other forms of IFNB-1a. Recent studies have reported a significant anti-inflammatory and neuroprotective effects of statins, cholesterol-lowering agents. Statins disrupt cellular membrane lipid rafts, which inhibit the clustering of T-cell receptor (TCR), co-stimulatory, and adhesion molecules, required for optimal T-cell activation. Along with inhibiting T-cell activation, statins decrease IFNB inducible MHC class II expression, suppressing an effective antigen presentation. They block migration of activated mononuclear cells from peripheral circulation into the CNS by blocking LFA-1 adhesion molecule and by reducing metalloproteinase type 9 secretion. While their anti-inflammatory effects at tolerable oral doses may not justify their use as monotherapy for RR MS, their pleiotropic mechanisms of action showed synergistic effects with IFNB-1a in studies in vitro. We propose that simvastatin may enhance the immunomodulatory effects of INFB-1a in patients with CIS suggestive of MS and that this combination may even more effectively prevent further disease activity if administered early in the course of the disease.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has a diagnosis of CIS suggestive of MS involving optic nerve (unilateral optic neuritis), spinal cord (incomplete transverse myelitis), brain stem or cerebellum syndrome confirmed by ophthalmologic or neurological examinations. (Onset of CIS symptoms must occur within twelve months of randomization).
2. At baseline, subject will be between the ages of 18 and 60, inclusive.
3. Subject has a baseline EDSS score between 0.0 and 5.5, inclusive.
4. MRI findings on the brain scan should reveal at least three out the four following findings: one Gd-enhancing lesion or nine T2 hyperintense lesions; or at least one infratentorial lesion; or at least one juxtacortical lesion and or at least three periventricular lesions.
5. Subject has signed informed consent and HIPAA forms.

Exclusion Criteria:

1. Subject has a diagnosis of CD RRMS according to Poser criteria, definitive MS according McDonald criteria, secondary progressive, or primary progressive MS.
2. Subject has been treated with statins in the previous three months. Subject has history of severe side effects related to statin therapy.
3. Subject has had a clinically significant infectious illness (e.g., cellulitis, abscess, pneumonia, septicemia) within 30 days prior to randomization.
4. Subject has a history of, or abnormal laboratory results indicative of, any significant cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, gastrointestinal, dermatologic, psychiatric, renal, and/or other major disease.
5. Subject has a history of severe allergic or anaphylactic reactions or known drug hypersensitivity.
6. Subject has an abnormal screening blood test, performed at the screening visit, exceeding any of the limits defined below:

   * alanine transaminase (ALT) or aspartate transaminase (AST) > 1.5 times the upper limit of normal (1.5x ULN)
   * total white blood cell count < 2,300/mm^3
   * CPK level > 2 x ULN on two consecutive occasions tested at least one week apart.
   * Platelets less than 150,00/mm3
   * Creatinine > 1.5mg/dl.
   * prothrombin time (PT) > ULN
7. Subject has history of treatment with either interferon-beta 1a or 1b, or glatiramer acetate.
8. Subject has had any prior treatment with any of the following medications:

   * total lymphoid irradiation
   * intravenous immunoglobulins IVIg, or plasma exchange
   * natalizumab or any other therapeutic monoclonal antibody
9. Subject has had treatment with any of the following medications within 1 year prior to randomization:

   * mitoxantrone
   * cyclophosphamide
10. Subject has had treatment with any of the following medications:

    * cyclosporine
    * azathioprine
    * methotrexate
    * glatiramer acetate
    * interferon beta-1b or INF beta-1a
    * intravenous immunoglobulin (IVIG)
    * plasmapheresis or cytapheresis
11. Subject has had treatment with any of the following medications within 50 days prior to randomization:

    * intravenous corticosteroid treatment
    * oral corticosteroid treatment
12. Subject has a history of alcohol abuse within 2 years prior to randomization.
13. Subject is a female who is not postmenopausal for at least one year, surgically sterile, or willing to practice effective contraception (as defined by the investigator) during the study. The rhythm method is not to be used as the sole method of contraception.
14. Subject is a nursing mother, pregnant woman, or planning to become pregnant while on study.
15. Subject has had participation in any other investigational study within 6 months prior to randomization.
16. Subject is unwilling or is unable to comply with the requirements of this protocol including the presence of any condition (physical, mental, or social) that is likely to affect the subject's ability to comply with the study protocol.
17. Subject is determined unsuitable for enrollment into this study for any other reason in the opinion of the Investigator and/or the Sponsor.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30
Dates: Start 2004-09; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to determine whether combination therapy with IFNb-1a plus simvastatin, when compared to IFNb-1a plus placebo decreases or delays additional clinical or MRI activity.
We will use the following outcome measures:
Relapse rates, Time to first relapse,Number of new T2 lesions, Number of new Gd-enhancing lesions

CONTACTS AND LOCATIONS:
Overall Officials: Silva Markovic-Plese, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina-Chapel Hill MS clinic within the Neuroscience Hospital, Chapel Hill, North Carolina, United States